CLINICAL TRIAL: NCT01739972
Title: Desiccated Thyroid Extract Compared to Levothyroxine in the Treatment of Hypothyroidism: A Randomized, Double-blind, Crossover Study.
Brief Title: Desiccated Thyroid Extract and Levothyroxine for Hypothyroidism Treatment
Acronym: DTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mohamed K.M. Shakir, Principal Investigator, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WalterReedNMMC
Record Dates: First submitted 2012-11-28; First posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Primary Hypothyroidism.
Keywords: Desiccated thyroid extract and levothyroxine
MeSH Terms: conditions — Hypothyroidism; Thyroid Diseases | interventions — Thyroxine; Thyroid (USP)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levothyroxine (Active Comparator): Levothyroxine in the capsule form, once daily, appropriate dosage to keep TSH at the normal range.
  Interventions: Drug: Desiccated thyroid extract
- Desiccated thyroid extract (Active Comparator): Desiccated thyroid extract in capsule form, once daily, appropriate dosage to keep TSH in the normal range.
  Interventions: Drug: Levothyroxine

INTERVENTIONS:
Drug: Levothyroxine — Levothyroxine in a capsule form, once daily, with appropriate dosage to keep TSH in the normal range.
  Other Names: Synthroid
  Arms: Desiccated thyroid extract
Drug: Desiccated thyroid extract — Armour thyroid in a capsule form, once daily, with appropriate dosage to keep TSH in normal range.
  Other Names: Armour Thyroid
  Arms: Levothyroxine

SUMMARY:
Our hypothesis is that hypothyroid patients on DTE may have a decrease in symptoms, an improvement of cognitive function, and an increase in sense of well-being/ quality of life equivalently compared with L-T4.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be between the ages of 18 to 65 and will have been on levothyroxine for primary hypothyroidism for at least 6 months.

Exclusion Criteria:

* Patients will be excluded if they have the following problems: pregnancy, plan for pregnancy in the next 12 months, cardiac disease, especially coronary artery disease, chronic obstructive lung disease, malabsorption disorder, gastrointestinal surgeries, significant renal or liver dysfunction, seizure disorders, thyroid and non-thyroid active cancers, uncontrolled psychosis, psychotropic medication use, steroid use, amiodarone, chemotherapy for cancer, iron supplement more than 325mg per day, carafate/ proton pump inhibitor use, cholestyramine use, and those with recent PCS orders who are expected to move out of the geographic area, age less than 18 years old or older than 65 years old.
* Patients scheduled for deployment will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
thyroid-symptom questionnaire | 4 months
  Thyroid Symptom Questionnaire, a health-related quality-of-life questionnaire, that consists of 12 questions, presented in the same format as the GHQ-12, that asked patients how they felt over the last three months.
Wechsler Memory Scale-Version IV (WMS-IV) | 4 months
  The Wechsler Memory Scale-Version IV (WMS-IV) included auditory memory index, visual memory index, visual working memory index, immediate memory index and delayed memory index.

SECONDARY OUTCOMES:
Biochemical measures | 4 months
  Biochemical testing consisting of serum TSH, free T4, total T4, total T3, T3 resin uptake, sex hormone binding globulin (SHBG), and a lipid panel.

OTHER OUTCOMES:
Beck Depression Index | 4 months
  The BDI is a self-rating scale of 21 items, in which scores of 10 or less indicate normal mood variation and scores of 11 or more reflect increasing levels of depression. Clinically important depression is associated with scores of 20 or more.
General health questionnaire-12 | 4 months
  General health questionnaire - consists of 12 quality of life questions.
Clinical preference | 4 months
  At the completion of the study, each patient will be asked which treatment (the first or the second) he or she preferred.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Walter Reed National Military Medical Center, Endocrinology, Bethesda, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland

REFERENCES:
- [Background] Roberts CG, Ladenson PW. Hypothyroidism. Lancet. 2004 Mar 6;363(9411):793-803. doi: 10.1016/S0140-6736(04)15696-1. PMID 15016491
- [Background] Cooper DS, Biondi B. Subclinical thyroid disease. Lancet. 2012 Mar 24;379(9821):1142-54. doi: 10.1016/S0140-6736(11)60276-6. Epub 2012 Jan 23. PMID 22273398
- [Background] Lowe JC. Stability, Effectivenes, and Safety of Desiccated Thyroid vs Levothyroxine: A Rebuttal to the British Thyroid Association. Thyroid Science 2009;4:C1-12.
- [Background] Sawin CT, Hershman JM, Fernandez-Garcia R, Ghazvinian S, Ganda OP, Azukizawa M. A comparison of thyroxine and desicatted thyroid in patients with primary hypothyroidism. Metabolism. 1978 Oct;27(10):1518-25. doi: 10.1016/s0026-0495(78)80024-9. No abstract available. PMID 99633
- [Background] Biondi B, Wartofsky L. Combination treatment with T4 and T3: toward personalized replacement therapy in hypothyroidism? J Clin Endocrinol Metab. 2012 Jul;97(7):2256-71. doi: 10.1210/jc.2011-3399. Epub 2012 May 16. PMID 22593590
- [Background] Celi FS, Zemskova M, Linderman JD, Smith S, Drinkard B, Sachdev V, Skarulis MC, Kozlosky M, Csako G, Costello R, Pucino F. Metabolic effects of liothyronine therapy in hypothyroidism: a randomized, double-blind, crossover trial of liothyronine versus levothyroxine. J Clin Endocrinol Metab. 2011 Nov;96(11):3466-74. doi: 10.1210/jc.2011-1329. Epub 2011 Aug 24. PMID 21865366
- [Background] Hennemann G, Docter R, Friesema EC, de Jong M, Krenning EP, Visser TJ. Plasma membrane transport of thyroid hormones and its role in thyroid hormone metabolism and bioavailability. Endocr Rev. 2001 Aug;22(4):451-76. doi: 10.1210/edrv.22.4.0435. PMID 11493579
- [Background] Salvatore D, Bartha T, Harney JW, Larsen PR. Molecular biological and biochemical characterization of the human type 2 selenodeiodinase. Endocrinology. 1996 Aug;137(8):3308-15. doi: 10.1210/endo.137.8.8754756.
- [Background] Kim BW, Bianco AC. For some, L-thyroxine replacement might not be enough: a genetic rationale. J Clin Endocrinol Metab. 2009 May;94(5):1521-3. doi: 10.1210/jc.2009-0410. No abstract available. PMID 19420275
- [Background] Panicker V, Saravanan P, Vaidya B, Evans J, Hattersley AT, Frayling TM, Dayan CM. Common variation in the DIO2 gene predicts baseline psychological well-being and response to combination thyroxine plus triiodothyronine therapy in hypothyroid patients. J Clin Endocrinol Metab. 2009 May;94(5):1623-9. doi: 10.1210/jc.2008-1301. Epub 2009 Feb 3. PMID 19190113
- [Background] Nygaard B, Jensen EW, Kvetny J, Jarlov A, Faber J. Effect of combination therapy with thyroxine (T4) and 3,5,3'-triiodothyronine versus T4 monotherapy in patients with hypothyroidism, a double-blind, randomised cross-over study. Eur J Endocrinol. 2009 Dec;161(6):895-902. doi: 10.1530/EJE-09-0542. Epub 2009 Aug 7. PMID 19666698
- [Background] Grozinsky-Glasberg S, Fraser A, Nahshoni E, Weizman A, Leibovici L. Thyroxine-triiodothyronine combination therapy versus thyroxine monotherapy for clinical hypothyroidism: meta-analysis of randomized controlled trials. J Clin Endocrinol Metab. 2006 Jul;91(7):2592-9. doi: 10.1210/jc.2006-0448. Epub 2006 May 2. PMID 16670166
- [Background] Escobar-Morreale HF, Botella-Carretero JI, Escobar del Rey F, Morreale de Escobar G. REVIEW: Treatment of hypothyroidism with combinations of levothyroxine plus liothyronine. J Clin Endocrinol Metab. 2005 Aug;90(8):4946-54. doi: 10.1210/jc.2005-0184. Epub 2005 May 31. PMID 15928247
- [Background] Appelhof BC, Fliers E, Wekking EM, Schene AH, Huyser J, Tijssen JG, Endert E, van Weert HC, Wiersinga WM. Combined therapy with levothyroxine and liothyronine in two ratios, compared with levothyroxine monotherapy in primary hypothyroidism: a double-blind, randomized, controlled clinical trial. J Clin Endocrinol Metab. 2005 May;90(5):2666-74. doi: 10.1210/jc.2004-2111. Epub 2005 Feb 10. PMID 15705921
- [Background] Saravanan P, Simmons DJ, Greenwood R, Peters TJ, Dayan CM. Partial substitution of thyroxine (T4) with tri-iodothyronine in patients on T4 replacement therapy: results of a large community-based randomized controlled trial. J Clin Endocrinol Metab. 2005 Feb;90(2):805-12. doi: 10.1210/jc.2004-1672. Epub 2004 Dec 7. PMID 15585551
- [Background] Escobar-Morreale HF, Botella-Carretero JI, Gomez-Bueno M, Galan JM, Barrios V, Sancho J. Thyroid hormone replacement therapy in primary hypothyroidism: a randomized trial comparing L-thyroxine plus liothyronine with L-thyroxine alone. Ann Intern Med. 2005 Mar 15;142(6):412-24. doi: 10.7326/0003-4819-142-6-200503150-00007. PMID 15767619
- [Background] Walsh JP, Shiels L, Lim EM, Bhagat CI, Ward LC, Stuckey BG, Dhaliwal SS, Chew GT, Bhagat MC, Cussons AJ. Combined thyroxine/liothyronine treatment does not improve well-being, quality of life, or cognitive function compared to thyroxine alone: a randomized controlled trial in patients with primary hypothyroidism. J Clin Endocrinol Metab. 2003 Oct;88(10):4543-50. doi: 10.1210/jc.2003-030249. PMID 14557419
- [Background] Clyde PW, Harari AE, Getka EJ, Shakir KM. Combined levothyroxine plus liothyronine compared with levothyroxine alone in primary hypothyroidism: a randomized controlled trial. JAMA. 2003 Dec 10;290(22):2952-8. doi: 10.1001/jama.290.22.2952. PMID 14665656
- [Background] Sawka AM, Gerstein HC, Marriott MJ, MacQueen GM, Joffe RT. Does a combination regimen of thyroxine (T4) and 3,5,3'-triiodothyronine improve depressive symptoms better than T4 alone in patients with hypothyroidism? Results of a double-blind, randomized, controlled trial. J Clin Endocrinol Metab. 2003 Oct;88(10):4551-5. doi: 10.1210/jc.2003-030139. PMID 14557420
- [Background] Bunevicius R, Kazanavicius G, Zalinkevicius R, Prange AJ Jr. Effects of thyroxine as compared with thyroxine plus triiodothyronine in patients with hypothyroidism. N Engl J Med. 1999 Feb 11;340(6):424-9. doi: 10.1056/NEJM199902113400603. PMID 9971866
- [Background] Bunevicius R, Prange AJ. Mental improvement after replacement therapy with thyroxine plus triiodothyronine: relationship to cause of hypothyroidism. Int J Neuropsychopharmacol. 2000 Jun;3(2):167-174. doi: 10.1017/S1461145700001826. PMID 11343593
- [Background] Smith RN, Taylor SA, Massey JC. Controlled clinical trial of combined triiodothyronine and thyroxine in the treatment of hypothyroidism. Br Med J. 1970 Oct 17;4(5728):145-8. doi: 10.1136/bmj.4.5728.145. PMID 4097650
- [Background] Lanni A, Moreno M, Lombardi A, Goglia F. Calorigenic effect of diiodothyronines in the rat. J Physiol. 1996 Aug 1;494 ( Pt 3)(Pt 3):831-7. doi: 10.1113/jphysiol.1996.sp021536. PMID 8865078
- [Background] Jackson IM, Cobb WE. Why does anyone still use desiccated thyroid USP? Am J Med. 1978 Feb;64(2):284-8. doi: 10.1016/0002-9343(78)90057-8. PMID 629277
- [Background] ROBERTSON JD, KIRKPATRICK HF. Changes in basal metabolism, serumprotein-bound iodine, and cholesterol during treatment of hypothyroidism with oral thyroid and L-thyroxine sodium. Br Med J. 1952 Mar 22;1(4759):624-8. doi: 10.1136/bmj.1.4759.624. No abstract available. PMID 14905006
- [Background] Means JH, Lerman J, Salter WT. THE ROLE OF THYROXIN IODINE AND TOTAL ORGANIC IODINE IN THE CALORIGENIC ACTION OF WHOLE THYROID GLAND. J Clin Invest. 1933 Jul;12(4):683-8. doi: 10.1172/JCI100529. No abstract available. PMID 16694154
- [Background] Thompson WO, McLellan LL, Thompson PK, Dickie LF. THE RATES OF UTILIZATION OF THYROXINE AND OF DESICCATED THYROID IN MAN: THE RELATION BETWEEN THE IODINE IN DESICCATED THYROID AND IN THYROXINE. J Clin Invest. 1933 Jan;12(1):235-46. doi: 10.1172/JCI100492. No abstract available. PMID 16694117
- [Background] Thompson WO, Thompson PK, Brailey AG, Cohen AC. THE CALORIGENETIC ACTION OF THYROXIN AT DIFFERENT LEVELS OF BASAL METABOLISM IN MYXEDEMA. J Clin Invest. 1929 Aug;7(3):437-63. doi: 10.1172/JCI100237. No abstract available. PMID 16693869
- [Background] McDowell I, Newell C. The General Health Questionnaire. Measuring Health. A Guide to Rating Scales and Questionnaires. 2nd Ed, Oxford, 1996
- [Background] Cooper DS, Halpern R, Wood LC, Levin AA, Ridgway EC. L-Thyroxine therapy in subclinical hypothyroidism. A double-blind, placebo-controlled trial. Ann Intern Med. 1984 Jul;101(1):18-24. doi: 10.7326/0003-4819-101-1-18. PMID 6428290
- [Background] Jaeschke R, Guyatt G, Cook D, Harper S, Gerstein HC. Spectrum of quality of life impairment in hypothyroidism. Qual Life Res. 1994 Oct;3(5):323-7. doi: 10.1007/BF00451724. PMID 7841966
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Benson N, Hulac DM, Kranzler JH. Independent examination of the Wechsler Adult Intelligence Scale-Fourth Edition (WAIS-IV): what does the WAIS-IV measure? Psychol Assess. 2010 Mar;22(1):121-30. doi: 10.1037/a0017767. PMID 20230158
- [Background] Wechsler DA. The Wechsler Memory Scale-III. 3rd ed. San Antonio, Tex:Psychological Corp;1997.